CLINICAL TRIAL: NCT04710017
Title: Tranexamic Acid Versus Depot-Medroxyprogesterone Acetate in the Treatment of Perimenopausal Irregular Uterine Bleeding: Randomized Clinical Trial
Brief Title: Tranexamic Acid and Depot-Medroxyprogesterone Acetate for Perimenopausal Irregular Uterine Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-DMPA
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Uterine Bleeding
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Tranexamic Acid; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid group (Other): will tranexamic acid 500 mg 4 times daily in one group,
  Interventions: Drug: Tranexamic acid
- Medroxyprogesterone acetate (Other): will receive 150mg of medroxyprogesterone acetate once intramuscular.
  Interventions: Drug: Medroxyprogesterone Acetate 150 MG/ML

INTERVENTIONS:
Drug: Tranexamic acid — will be given Tranexamic acid at 500 mg four times daily (2 g/day) during the bleeding episodes for 5 days. The dose is 250 mg.
  Arms: Tranexamic acid group
Drug: Medroxyprogesterone Acetate 150 MG/ML — will be given MPA at 150 mg once intramuscular injection
  Arms: Medroxyprogesterone acetate

SUMMARY:
Abnormal uterine bleeding is a symptom and not a disease. It is one of the most frequently encountered complaints in gynecologic practice. It accounts for more than 70% of all gynecological consultations in the peri- and post-menopausal age group.

Abnormal uterine bleeding may be acute or chronic and is defined as bleeding from the uterine corpus that is abnormal in regularity, volume, frequency, or duration and occurs in the absence of pregnancy.

Chronic heavy or prolonged uterine bleeding can result in anemia, interfere with daily activities. Iron deficiency anemia develops in 21 to 67 percent of cases and raises concerns about uterine cancer.

According to the International Federation of Obstetrics and Gynecology, the classification of abnormal uterine bleeding is based on PALM-COEIN which is an acronym for various etiologies namely polyp, adenomyosis, leiomyoma, malignancy and hyperplasia, coagulopathy, ovulatory dysfunction, endometrial disorders, iatrogenic and not otherwise classified (PALM-COEIN).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed, clinically as peri-menopausal abnormal uterine bleeding with normal pelvic examination.
* Patient's age ranging from 40- 55y.

Exclusion Criteria:

* Post menopausal women
* Presence of fibroids, adenomyosis, polyp, adnexal mass, endometrial hyperplasia with atypia, and breast malignancy).
* Patients with uncontrolled hypertension.
* Patient of abnormal bleeding profile.
* history of liver impairment and renal insufficiency
* Patients seeking for surgical management.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Number of bleeding days | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided